CLINICAL TRIAL: NCT05255185
Title: Can "Domino" Therapy Effectively Treat the Infection Around the Prosthesis After the Limb Salvage Surgery of Bone Tumor？-----A Study of Sequential Therapy
Brief Title: "Domino" Therapy Treat the Infection Around the Prosthesis After the Limb Salvage Surgery of Bone Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0151
Record Dates: First submitted 2022-01-25; First posted 2022-02-24 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-01

CONDITIONS: Infection
Keywords: Bone tumor; Limb salvage surgery; infection; Therapy effect
MeSH Terms: conditions — Infections; Bone Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All the patients (Experimental): domino therapy treat the infection around the prosthesis after the limb salvage surgery of bone tumor
  Interventions: Procedure: domino therapy

INTERVENTIONS:
Procedure: domino therapy — The investigators evaluated routine blood test results, C-reactive protein level, the erythrocyte sedimentation rate, and other indicators. X-rays and CT scans of the surgical site were obtained and the Musculoskeletal Tumor Society (MSTS) score was calculated. Treatment involved debridement and lavage of the prosthesis, and systemic and local antibiotics.

SUMMARY:
Tumor resection and prosthetic replacement have become the treatments of choice for malignant bone tumors. Infections are the main cause of failure of limb salvage surgeries. Therefore, treatment of infections around prostheses after limb salvage is important, but is also challenging. Our research team designed a "domino" sequential treatment plan to treat postoperative infections around tumor prostheses and evaluated its efficacy.

DETAILED DESCRIPTION:
Malignant bone tumors are associated with high mortality and disability rates. Developments over the past 20 years have made tumor resection and prosthetic replacement the preferred surgical treatments. Prosthetic reconstruction maintains the continuity of limb bones and leads to better joint function, but is often associated with complications such as loosening, fracture, and infection of the prosthesis. Among these, infection is the most important cause of failed limb salvage surgery. Postoperative infection rates of 5-25% have been reported in the literature. Infection is also the main cause of secondary amputation. Therefore, it is important to address infections around the prosthesis after limb salvage.

Investigators retrospectively analyzed the use of prosthesis-preserving sequential therapy to treat patients with peripheral prosthesis infections after bone-tumor limb salvage. Investigators summarized and analyzed the treatment processes and performed laboratory, imaging, and functional evaluations after treatment. The purpose was to introduce a new type of domino sequential treatment plan for treating postoperative infections of tumor prosthesis, and evaluate the technical points of the plan, and prognosis over medium- and long-term follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Deep postoperative infections after replacement of a tumor-type prosthesis according to the 2011 diagnostic criteria of the Musculoskeletal Infection Society (MSIS) ;
* Treated with debridement and lavage with prosthesis preservation, local application of antibiotics, and no loosening during intraoperative exploration;
* With complete data for the main indicators (routine blood test results, C-reactive protein [CRP] level, erythrocyte sedimentation rate [ESR], X-ray and CT scans of the surgical site, and the Musculoskeletal Tumor Society [MTST] score).

Exclusion Criteria:

* Underwent debridement without prosthesis preservation;
* With a loose prosthesis during intraoperative exploration;
* With poor soft tissue coverage, such that complete free muscle flap coverage could not be achieved; patients with renal insufficiency/failure (serum creatinine ≥ 2.0 mg/dL); patients with uncontrolled diabetes mellitus (hemoglobin A1c level > 8%);
* In poor general condition who could not tolerate surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
success rate of patients undergoing domino therapy assessed by MSIS diagnostic criteria | 4 years
  Sequential treatment failure was defined as failure to treat infection within 2 years of follow-up, indicated by meeting the 2011 MSIS diagnostic criteria of infection around the prosthesis.
  The following formula was used to calculate the success rate: success rate = (total number of patients-number of failed cases)/total number of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoming Ye, Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Department of Orthopedics, The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China